CLINICAL TRIAL: NCT04167540
Title: Open-Label Safety Study of Glial Cell Line-Derived Neurotrophic Factor Gene Transfer (AAV2- GDNF) in Parkinson's Disease
Brief Title: GDNF Gene Therapy for Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brain Neurotherapy Bio, Inc. (Industry)
Collaborators: AskBio Inc (Industry); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDNF-102
Record Dates: First submitted 2019-11-07; First posted 2019-11-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease
Keywords: PD; Parkinson's disease; Neurotrophic factor; Growth factor; Glial cell line-derived neurotrophic factor; GDNF; AAV; Gene therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A total of 12 study participants will be administered the investigational product in this Phase 1b trial. Participants will be enrolled into cohorts, based upon the duration and stage of their PD. Six (6) participants will be dosed in each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Earlier stage PD (Experimental)
  Interventions: Biological: AAV2-GDNF
- Later stage PD (Experimental)
  Interventions: Biological: AAV2-GDNF

INTERVENTIONS:
Biological: AAV2-GDNF — Bilateral image-guided infusion of AAV2-GDNF into putamen, single dose

SUMMARY:
The objective of this Phase 1b investigation is to evaluate the safety and potential clinical effect of AAV2-GDNF delivered to the putamen in subjects with either a recent or a long-standing diagnosis of PD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female adults 35-75 years of age (inclusive)
* Diagnosed with Parkinson's disease
* Modified Hoehn and Yahr stage I-III OFF medication
* Time since receiving a clinical diagnosis of PD and disease severity consistent with one of the following:

  1. EITHER: Less than 5 years since clinical diagnosis of PD and mild to moderate UPDRS III OFF score
  2. OR: At least 4 years since clinical diagnosis of PD and moderate to severe UPDRS III OFF score
* Responsiveness to levodopa

Key Exclusion Criteria:

* Atypical parkinsonism
* Severe dyskinesia
* Presence of dementia, psychosis, substance abuse or qualify as "severe depression"
* Prior brain surgery (i.e. deep brain stimulator or DBS implantation) or other brain imaging abnormalities
* Receiving an investigational drug
* History of cancer or poorly controlled medical conditions that would increase surgical risk
* Inability to tolerate laying flat in an MRI or allergy to gadolinium

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of Treatment-Emergent Adverse Events (TEAE) assessed clinically by physical and neurological examinations | 5 years
  Evaluation of the safety and tolerability through the assessment of incidence of TEAE, identified by MedDRA preferred term and grouped by MedDRA System Organ Class, as well as clinically meaningful changes in clinical exams or laboratory assays.

SECONDARY OUTCOMES:
Motor symptoms as assessed by the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 18 months
  Change from baseline in the MDS-UPDRS. The MDS-UPDRS contains 4 subscales: Part I, non-motor aspects of experiences of daily living (13 items); Part II, motor aspects of experiences of daily living (13 items); Part III, motor examination (33 scores based on 18 items); Part IV, motor complications (6 items). The rating for each item, or sub-item, is from 0 (normal) to 4 (severe). The total score for each Part is obtained from the sum of the corresponding item scores.
Non-motor symptoms of Parkinson's disease as assessed by the Non-Motor Symptom Scale (NMSS) | 18 months
  Change from baseline in the NMSS. The NMSS evaluates 9 domains of non-motor of severity and frequency of PD symptoms associated with cardiovascular health, sleep and fatigue, mood and cognition, perceptual problems and hallucinations, attention and memory, gastrointestinal tract, urinary, sexual function, and a miscellaneous domain for other common non-motor conditions. Severity x frequency scores range 0-108, with 0 being less severe and less frequent.
Brain dopaminergic cell integrity as measured by DaTscan | 18 months
  Percentage and absolute changes in Ioflupane retention as a marker for dopamine transporter protein expressed by dopamine producing cells within the brain. Measured by quantitative analysis of DaTscan SPECT imaging.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Irvine, Irvine, California
  - University of California San Francisco, San Francisco, California
  - The Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No